CLINICAL TRIAL: NCT03973060
Title: Effectiveness of Muscular Work in Strength Gain of Ischiofemoral and Quadriceps: Relationshionship of Genetic Variants in Improvement of Explosive Force
Brief Title: Effectiveness of Muscular Work and Genetic Variants in Strength Gain of Ischiofemoral and Quadriceps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Collaborators: Sofía Laguarta Val (Unknown); Alberto Melián Ortiz (Unknown)
Responsible Party: Principal Investigator, David Varillas Delgado, Research Unit Director, Universidad Francisco de Vitoria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URJC
Record Dates: First submitted 2019-05-28; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Muscle Strength; Genetics
Keywords: Jump test; Genetic polymorphism; Muscle strength; Physiotherapies techniques
MeSH Terms: interventions — Polymorphism, Genetic; Dipeptidyl-Peptidases and Tripeptidyl-Peptidases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant was blinded not knowing the treatment to which he was submitted and outcome assessor responsible for collecting the results, without commenting on the group from which the patient came. Only the principal investigator knew the group to which the patient belonged.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Concentric muscular work (Experimental): 4 series of 12 repetitions of concentric muscular work, with one minute rest between each repetitions, total working time of 24 minutes.
  Interventions: Device: Concentric-eccentric muscular work; Genetic: Genetic polymorphism
- Eccentric muscular work (Experimental): 4 series of 12 repetitions of eccentric muscular work, with one minute rest between each repetitions, total working time of 24 minutes.
  Interventions: Device: Concentric-eccentric muscular work; Genetic: Genetic polymorphism
- Concentric-eccentric muscular work (Experimental): 4 series of 12 repetitions of concentric-eccentric muscular work, with one minute rest between each repetitions, total working time of 24 minutes.
  Interventions: Device: Concentric-eccentric muscular work; Genetic: Genetic polymorphism
- Isometric muscular work (Experimental): 6 seconds of contraction, with 20 seconds of rest with 24 repetitions, for a total working time of 12 minutes.
  Interventions: Device: Concentric-eccentric muscular work; Genetic: Genetic polymorphism

INTERVENTIONS:
Device: Concentric-eccentric muscular work — For muscular contraction, the physiotherapist carried out 12 repetitions with one minute rest between series and series, total working time of 12 minutes.
  Other Names: Muscular work; Vertical jump; 60m sprint; Jump potence; Horizontal jump
Genetic: Genetic polymorphism — Genetic polymorphism study by Polymerase Chain Reaction (PCR) to determine whether the genetic makeup of individuals for the improvement of muscular work in the results of the study.
  Other Names: ACTN3 gene; ACE gene

SUMMARY:
In the field of sports training and recovery, the work of muscular strength has become the star theme in terms of its influence on the performance of athletes. In fact, in relation to the training of the inferior members, the scientific evidence indicates that, to increase the other two physical qualities conditioned (speed and resistance), it is necessary to work and to increase the muscular strength.

Randomized intervention trial with sample size of 80 subjects divided into 4 groups (n = 20) of muscular work: concentric, eccentric, concentric-eccentric and isometric. Ages between 21-23 years.

For all the above, the investigators will study as a main objective analyze what type of muscular work is most effective in order to improve some variables of the performance of explosive muscular strength, and to try to determine if that improvement is due, exclusively to the developed training or to the genetics of the subjects and compare the results obtained in the variables of vertical jump, power of saint, horizontal jump and speed 60 meters, before and after the execution of each one of the muscular works dynamic among themselves, and compared to the muscular work isometric.

DETAILED DESCRIPTION:
In the field of sports training and recovery, the work of muscular strength has become the star theme in terms of its influence on the performance of athletes. In fact, in relation to the training of the inferior members, the scientific evidence indicates that, to increase the other two physical qualities conditioned (speed and resistance), it is necessary to work and to increase the muscular strength.

To this end, numerous training methods have been developed, in which research and technology provide new solutions that favor and enhance the muscular work done.

Therefore, in the performance of an athlete this work of force influences, and what this implies: type of muscular contraction, way of working that contraction, recruitment of the muscular fiber, and modality of muscular strength developed. But, this performance, it appears that it can also be influenced by environmental parameters such as diet, technological support and genetic factors. It has been discovered in the human genome 12 million of polymorphisms, but it is only recorded that some 214 may have influence on physical qualities, and all of them, the most studied in terms of their influence on sports performance are: genes Muscular, and more specifically the ACTN3, and vasomotor genes that affect the production of energy and that intervene in metabolic processes (ACE gene).

* Design: Randomized intervention clinical trial, double blinded.
* Sample: by contrast of hypothesis, a sample size of 80 subjects divided into 4 groups (n = 20) of muscular work: concentric, eccentric, concentric-eccentric and isometric. They were randomized using excel software. As criteria of inclusion, subjects that did not present musculoskeletal lesions in the lower train at the time of the study, which showed a serious commitment to perform the entire muscle training, which were not subject to another type of plan Training that could interfere with the results obtained from the measurement of the study variables, and that would not have been diagnosed with hypertension.
* Methodology:

The duration of the muscular work was 12 consecutive days, measuring before and after the same variables indicated below.

The protocol of work was as follows: 4 series of 12 repetitions of the type of muscular contraction of each group, with one minute of rest between series and series. For the muscular work isometric: 6 seconds of contraction, with 20 seconds of rest, for a total working time of 12 minutes.

As a material for muscular work, the muscle brace or Russian belt was used for the three types of dynamic muscular work and the quadriceps bench for isometric muscular work. Other variables that were taken into account were: sex, age, weight, height, body mass index, blood pressure and heart rate.

As explosive force variables were measured: The Jump Power (Sayers formula), the vertical jump (the Sargent jump test), horizontal jump and speed 60 meters.

Other variables that were taken into account were: sex, age, weight, height, body mass index, blood pressure and heart rate.

At the end of the 12 days of training was extracted 10 ml of blood to each subject of the sample, then obtain the DNA analysis of the genotypes of the two genes analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that did not present musculoskeletal lesions in the lower train at the time of the study.
* Subjects that showed a serious commitment to perform the entire muscle training.
* Subjects not subject to another type of training plan that could interfere with the results obtained from the measurement of the study variables.

Exclusion Criteria:

* Subjects with high blood pressure.

Ages: 21 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
Jump power | Changes from baseline and at the end of procedure (12 days)
  Mechanical power in jump tests were measured by estimated (indirect way) from a subject's jump height and body mass, by means of Sayers equation.
Vertical jump | Changes from baseline and at the end of procedure (12 days)
  The protocol followed for the measurement was; First time: When the patient was barefoot, he placed himself sideways to a smooth wall and raised his right arm with his hand flat on the wall; The distance from the ground to the third finger of the hand (H1) was then measured. Second time: The subject was impregnated the third finger of the right hand in blue chalk powder, separated 10 centimeters from the wall and made a jump back movement with freedom to flex the lower limbs to the 90 º and move the arms, to consecutively and without any pause make a maximum vertical jump. Subsequently, this new distance was measured. This jump was made three times with a break between jump and jump of 45 seconds, and the average of the three (H2) was obtained. Third time: The value of the vertical jump was H = h1-h2.
Horizontal jump | Changes from baseline and at the end of procedure (12 days)
  On a smooth and horizontal surface, different marks were made distanced one meter each. In the first mark the subject was placed with the feet slightly separated at the height of the hips. Then a first test jump was made; To do so, the subject was told to swing with his arms and bending his knees, he had to jump forward with the greatest possible power. Once this first Test jump was made, the second measurement was carried out, the result of which was taken into account. This result was obtained in centimeters by means of measuring tape, with a precision of one millimeter (mm), and having as points of reference the first mark and the heel of the foot more retarded. The jump was not valid if the first mark was exceeded with the feet before taking off from the ground.
60 meters sprint | Changes from baseline and at the end of procedure (12 days)
  On an unobstructed sand surface, a distance of 60 meters was pointed out. The measurement in seconds of this variable was obtained by means of a stopwatch.

SECONDARY OUTCOMES:
ACTN3 polymorphism | Baseline.
  Blood sample was taken from 10ml in EDTA tube to all subjects in the study and by PCR analyzed the polymorphism R577X which is defined in the bibliography as a predetermined for the type of muscle fibers.
ACE polymorphism | Baseline.
  Blood sample was taken from 10ml in EDTA tube to all subjects in the study and by PCR analyzed the polymorphism I/D that is defined in the bibliography as influential in blood pressure.

OTHER OUTCOMES:
Cardiac frequency | Changes from baseline and at the end of procedure (12 days).
  Analyze cardiac frequence modifications in each intervention groups previous procedure, during the procedure and at the end of procedure.
Systolic and Diastolic blood pressure | Changes from baseline and at the end of procedure (12 days).
  Analyze both blood pressures (systolic and diastolic) modifications in each intervention groups previous procedure, during the procedure and at the end of procedure.